CLINICAL TRIAL: NCT04435249
Title: Phase I/II, Open Label Study to Assess the Safety and Efficacy Autologous Bone Marrow-derived Mesenchymal Stromal Cells Seeded on to Decellularised Airway Scaffold in Subjects with Clinically Significant Bronchopleural Fistula
Brief Title: ENgineered Tissue Repair of BronchopleUral FiSTula
Acronym: ENTRUST
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding constraints
Sponsor: Videregen Limited (Industry)
Collaborators: Cell Therapy Catapult (Other); Papworth Hospital NHS Foundation Trust (Other Government); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UK-2019-004939-24
Record Dates: First submitted 2020-05-29; First posted 2020-06-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Bronchopleural Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Patients will have a patch of expanded somatic mesenchymal stromal cells (MSCs) seeded onto a decellularised human tracheal-scaffold surgically implanted to repair bronchial fistula.
  Interventions: Other: BPF-001

INTERVENTIONS:
Other: BPF-001 — Expanded somatic mesenchymal stromal cells (MSCs) seeded onto a decellularised human tracheal-scaffold

SUMMARY:
Phase I/II Open-label Study to Assess the Safety and Efficacy of a Novel Tissue Engineered Airway Product, Consisting of Expanded Autologous Bone Marrow (BM) Derived Mesenchymal Stromal Cells (MSC) Seeded on to a Decellularised Allogeneic Patch of an Airway Scaffold in Subjects With Clinically Significant Bronchopleural Fistula.

DETAILED DESCRIPTION:
The proposed clinical trial is a phase I/II open-label study to assess the safety and efficacy of a novel tissue engineered airway product, consisting of expanded autologous Bone Marrow (BM) derived Mesenchymal Stromal Cells (MSC) seeded on to a decellularised allogeneic patch of an airway scaffold in subjects with clinically significant bronchopleural fistula. It is a phase I/II open-label study, which is an uncontrolled pilot in 5 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years or older.
* Documented diagnoses of BPF through imaging and bronchoscopic examination.
* BPF which involves the tracheobronchial junction or proximal bronchus.
* Subjects who have failed primary repair.
* Subjects who have no evidence of any primary or recurrent cancer (not limited to the surgical site) at the time of pre-operative screening as evidenced by CT and/or targeted biopsy (except for controlled or controllable basal cell carcinoma.
* Subjects who have signed and dated written informed consent to participate in the study.
* Females of childbearing potential (i.e. not surgically sterilised or post-menopausal for at least 2 years) must have a negative serum or urine pregnancy test.
* Male and female subjects of childbearing potential (i.e. not surgically sterilised or post-menopausal for at least 2 years) must use forms of highly effective methods of contraception, which are defined as hormonal methods of contraception (oral, injection or implant), barrier methods (condom or occlusive cap (diaphragm or cervical/vault caps)) with spermicidal foam/gel/cream/film/suppository, or true abstinence for 1 month following surgery.
* Subjects who have produced viable cells from Bone Marrow Aspirate.

Exclusion Criteria:

* Subjects who have received previous treatment with another Advanced Technology Medicinal Product (ATMP).
* Subjects with ECOG performance status of 3 or 4.
* Subjects deemed not suitable for surgery by the MDT.
* Uncontrolled diabetes, defined as HbA1c levels above 7.0 %.
* Any medical condition contraindicating the ability to tolerate general anaesthetic in the judgement of a consultant anaesthetist.
* Subjects who have a severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
* Subjects with clinically significant renal and liver impairment.
* Subjects undergoing an immunosuppression regimen or suffering from a primary immunodeficiency syndrome.
* Subjects with any known hypersensitivity to the culture and transport media compounds.
* Subjects with current or recurrent disease that could affect the administration, the action or disposition of the investigational product, or clinical or laboratory assessments.
* Subjects with clinically relevant or recent (within 2 years) history of substance abuse, including alcohol.
* Subject who has participated in any other interventional clinical trial within previous 30 days of the start of this study.
* Subjects with known presence of Human Immunodeficiency Virus (HIV) antibody, Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody.
* Subject who, in the investigator's judgement, is unlikely to complete all protocol required study visits or procedures, including follow-up visits, or comply with the study requirements for participation
* Subjects with any medical condition, that in the investigator's judgement, is likely to interfere with assessment of safety or efficacy of study treatment.
* Subject who is pregnant.
* Subjects with cancer (except for controlled or controllable basal cell carcinoma).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Safety: Emergent or worsening Serious Adverse Events (SAEs) related to the BPF implant during the 3 months post-defect repair | 3 months (90 days)
  Safety: Emergent or worsening Serious Adverse Events (SAEs) related to the BPF implant during the 3 months post-defect repair.
Efficacy: Bronchopleural Fistula (BPF) closure at 3 months assessed by visual appearance and no clinical signs of leaks. | 3 months (90 days)
  Closure of BPF with no need for further surgical closure. Efficacy will be deemed demonstrated if 2 or more subjects meet the primary endpoint.

SECONDARY OUTCOMES:
Change from Baseline in Physiological and Quality of Life scores at 3, 6, 9, 12 months, Evaluation Questionnaire 5D (EQ-5D), 6-minute walking test (6MWT), ambulatory oxygen (O2). | 36 months
  Impact as assessed in change from Baseline in Physiological and Quality of Life scores for each subject at 3, 6, 9, 12, 24 and up to 36 months post defect repair: QoL EQ-5D, 6-minute walking test, ambulatory O2 measurements.
Safety and tolerability: - Adverse Events (AEs) including pre-defined postoperative AEs of special interest up to 30± 3 days post implantation- Related AEs reported after 3, 6, 9, 12, 24 and 36 months | 36 months
  Adverse events related to the BPF implant procedures reported after 3, 6, 9, 12, 24 and 36 months.
Viability and the integrity of the repair area (closure) visually via bronchoscope. Integrity assessed by visual appearance of no visible leaks- Structural closure of the defect and visual health of the defect area and surrounding tissue | 36 months
  viability of the repair area and integration with vascular supply at 6, 9, 12, 24 and 36 months.
Absence of other surgical interventions at 6, 9, 12, 24 and 36 months | 36 months
  Interventions at the operative sites up to 6, 9, 12, 24 and 36 months

IPD SHARING:
Plan to Share IPD: No
to follow